CLINICAL TRIAL: NCT03692663
Title: Clinical Study on the Safety and Efficacy of Anti-PSMA CAR NK Cells in Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Study of Anti-PSMA CAR NK Cell (TABP EIC) in Metastatic Castration-Resistant Prostate Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Collaborators: Tianjin People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TABP EIC-01
Record Dates: First submitted 2018-09-29; First posted 2018-10-02 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TABP EIC treatment group (Experimental): Drug: TABP EIC Experimental Interventional Therapy
  Interventions: Drug: TABP EIC; Biological: Cyclophosphamide; Biological: fludarabine

INTERVENTIONS:
Drug: TABP EIC — A single dose of 0.5, 10, and 30 million TABP EIC will be iv administered at D0, D7, and D14.
Biological: Cyclophosphamide — Cyclophosphamide will be iv administered with 250 mg/m^2 at D-3, D-2, and D-1 before TABP EIC infusion.
Biological: fludarabine — Fludarabine will be iv administered with 25 mg/m^2 at D-3, D-2, and D-1 before TABP EIC infusion.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and preliminary efficacy of TABP EIC in patients with Metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

To enter the trial, subjects had to meet all of the following eligibility criteria:

1. diagnosed metastatic castration-resistant prostate cancer (mCRPC);
2. Castration level of serum testosterone (< 50 ng/dL or < 1.7 nmol/L);
3. Positive expression of PSMA;
4. According to the definition of CRPC in the Guidelines for the Diagnosis and Treatment of Prostate Cancer (2022 edition), the disease still progresses after castration and meets any of the following criteria:

   A.According to the increase in PSA level, there should be 3 consecutive increases in PSA at least 1 week apart (the increase in PSA is more than 50% of the minimum value, and PSA > 2 ng/mL); B.Progression of bone disease as defined by PCWG3, defined as the presence of 2 or more new lesions on bone scan; C.CT or MRI results suggested measurable metastasis (lymph node short diameter > 15 mm was defined as lymph node metastasis as assessed by RECIST 1.1);
5. Expected survival time ≥6 months;
6. Toxicity of any previous treatment had recovered to ≤ grade 1 at the time of enrollment (except hair loss and hearing loss);
7. ECOG score of patients 0-1;
8. Patients voluntarily participated and signed the informed consent, and followed the trial treatment plan and visit plan.

Exclusion Criteria:

Subjects who meet one of the following conditions will not be enrolled in the trial:

1. Previous recipients of other cell therapy products, such as dendritic cells (DC), multiple cytokine-induced killer cells (CIK), T cells, natural killer cells (NK), chimeric antigen receptor T-cell immunotherapy (CAR-T), etc.;
2. Previous treatment with any PSMA-targeted therapy;
3. radiotherapy was administered within 4 weeks prior to the start of study treatment;
4. Patients with a history of biological macromolecule drug allergy;
5. Abnormal function of major organs:

   A. Neutrophil count (ANC) < 1.5×109/L; Platelet count (Plt) < 100×109/L; Hemoglobin (Hb) < 9 g/dL; B. Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥2.5×ULN (≥5×ULN for liver metastases); C. Renal function: serum creatinine (Cr) ≥1.5×ULN; D. Prothrombin time (PT) > 15 s, activated partial thrombin time (APTT) was prolonged or shortened by more than 10 s (normal reference value 23 s-37 s), or international normalized ratio (INR) > 1.7; E. Pulmonary function: Severe respiratory diseases (active pulmonary tuberculosis, chronic obstructive pulmonary disease, interstitial lung disease, etc.)
6. Patients required systemic long-term steroid use or had received systemic steroids (dose equivalent to prednisone >10 mg/ day, except for patients using inhaled hormones) or other immunosuppressive agents 30 days before enrollment;
7. A history of severe central nervous system disorders, such as stroke or epilepsy;
8. active autoimmune diseases (including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease, or multiple sclerosis) or need long-term immunosuppressive therapy of severe autoimmune disease (screening clinic within six weeks before any immunosuppressive therapy), or by the researchers determine in 3 months will be recurrence of subjects;
9. have had other malignancies other than prostate cancer (other than basal or squamous cell skin cancer) in the past 5 years that are currently clinically significant and require intervention;
10. Clinically significant heart disease (New York Heart Association class III/IV, left ventricular ejection fraction < 60%);
11. Any active (viral, bacterial, fungal) infection currently being treated or any infection requiring intravenous antibiotics for 7 or more days or intervals during the past 6 weeks or any active infection requiring oral antibiotics during the past 1 week;
12. untreated chronic active hepatitis B, or chronic hepatitis B virus carriers with HBV DNA≥1000 copies /mL, or active hepatitis C patients;
13. Patients who have participated in other clinical trials and used study drugs within 3 months;
14. In the opinion of the investigator, there are other factors that are not suitable for inclusion or affect the participant's participation or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events as assessed by CTCAE v5.0 | Baseline to 1 year post infusion
  Defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
The pharmacokinetic analysis of TABP EIC | D0, D1, D3, D7, D8, D10, D14, D15, D17, D28±1, D60±2, D120±2, D180±7, D270±7, and D365±7 post infusion
  Changes in the number of CD56+/ CD3-TABP EIC in peripheral blood over time
The pharmacodynamics analysis of TABP EIC | Baseline to infusion date, D28±1, D60±2, D120±2, D180±7, D270±7, 和 D365±7
  Changes of total prostate specific antigen (tPSA) and free prostate specific antigen (fPSA) in peripheral blood
The proportion of patients with a decrease in PSA levels from baseline. | Baseline to D28±1, D60±2, D120±2, D180±7, D270±7, and D365±7 post infusion
  PSA response rate
Progression-free survival (PFS) after TABPEIC infusion | Baseline to 1 year post infusion
  Survival time of patients
Time to clinical progression | Baseline to D28±1, D60±2, D120±2, D180±7, D270±7, and D365±7 post infusion
  The time from baseline to the appearance of increased PSA levels or imaging progression.

CONTACTS AND LOCATIONS:
Overall Officials: Huaqing Wang, Doctor, Principal Investigator — Oncology of Tianjin people's hospital, 190 Jianyuan Road, Hongqiao District, Tianjin; Jian Li, Doctor, Principal Investigator — Urinary surgeryof Tianjin people's hospital, 190 Jianyuan Road, Hongqiao District, Tianjin
Locations (1):
- Tianjin pepole's hosptial, Tianjin, China

IPD SHARING:
Plan to Share IPD: No